CLINICAL TRIAL: NCT03469518
Title: Systemic and Intestinal Therapeutic Target Bioactivity of a Functional Beverage Containing β-cryptoxanthin (β-Cx), Plant Sterols (PS) and Galactooligosaccharides (GOS): "in Vivo" and "in Vitro" Studies.
Brief Title: Effect of β-cryptoxanthin (β-Cx), Plant Sterols and Galactooligosaccharides on Systemic and Gastrointestinal Markers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Nutrition and Food Science Area, Faculty of Pharmacy, University of Valencia (Unknown); Global Technology centro, Hero Group (Unknown); Fundación para la Investigación Biomédica, Hospital Universitario Puerta de Hierro (Unknown)
Responsible Party: Principal Investigator, Fernando Granado Lorencio, Principal Investigator. Chief Assistance., Puerta de Hierro University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AGL2015-68006-C2-2-R
Record Dates: First submitted 2018-02-19; First posted 2018-03-19 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Hypercholesterolemia; Osteoporosis; Postmenopausal Disorder
Keywords: beta-cryptoxanthin; cholesterol; Galactooligosaccharides; Plant Sterols; Cardiovascular risk; Bone Turnover markers; Intestinal Inflammatory markers; Microbiota
MeSH Terms: conditions — Hypercholesterolemia; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Crossover Assigment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-Cx plus PS (Sham Comparator): Fruit and milk based beverage enriched with beta-cryptoxanthin and plant sterols
  Interventions: Dietary Supplement: β-Cx plus PS
- β-Cx plus PS plus GOS (Active Comparator): Fruit and milk bases beverage enriched with beta-criptoxanthin, plant sterols and galactooligosaccharides
  Interventions: Dietary Supplement: β-Cx plus PS plus GOS

INTERVENTIONS:
Dietary Supplement: β-Cx plus PS plus GOS
  Arms: β-Cx plus PS plus GOS
Dietary Supplement: β-Cx plus PS
  Arms: β-Cx plus PS

SUMMARY:
Regular consumption of a beverage containing β-cryptoxanthin (β-Cx) and plant sterols (PS) has been shown to exert a synergic effect in reducing some markers of cardiovascular risk and bone-remodeling (formation and resorption). The present project aims to:

* Evaluate (by in vivo and in vitro studies) the bioavailability of added β-Cx, PS and galactooligosaccharides (GOS) and its stability in the beverage employed in the proposed study.
* Study the biological effect (bioefficacy) associated with the regular consumption of modified milk-based fruit beverages containing β-Cx, PS and GOS in post-menopausal women (target group) by assessing changes in inflammation, cardiovascular and bone turnover biochemical markers.
* Characterize genetic variability (polymorphisms), genetic expression and DNA oxidative damage in the target group as determinants of bioavailability and biological effects of β-Cx, PS and GOS.
* Evaluate the potential prebiotic effect associated to regular consumption of a beverage supplemented with β-Cx, PS and GOS: including "in vitro" studies and characterization of subjects' microbiota and possible microbiota changes associated to the beverage consumption.

DETAILED DESCRIPTION:
A previous Clinical Trial (AGL2012-39503-C02) evidenced the beneficial synergic effects upon bone remodeling and cardiovascular risk of a beverage, based on juice and milk, and enriched with PS and β-Cx. "In vitro" and "in vivo" (clinical) studies have confirmed low absorption of PS and β-Cx in this beverage, with possible slight modification of the sterols and metabolites by the intestinal microbiota. PS and β-Cx can reach the colon and be transformed by the intestinal microbiota with resulting beneficial effects.

The new Clinical Trial aims to determine whether the presence of galactooligosaccharides (GOS) in a beverage containing PS and β-Cx might modulate the biological effects of these latter components at either intestinal level (modification of microbiota and inflammatory markers) or systemically (blood cholesterol-lowering effect and bone turnover).

In the present clinical interventional study we will evaluate the systemic biological effects of a beverage containing GOS, PS and β-Cx, as well as its intestinal effects and its influence on the microbiota in postmenopausal women. Furthermore, we will study the stability and bioavailability of PS and β-Cx in the beverage.

The clinical study will help to confirm whether the new GOS-containing beverage has effects upon cardiovascular risk markers, bone remodeling and inflammation at least equivalent to those observed with the beverage studied in the previous Clinical Trial.

The results obtained will generate interesting information for improving beverage formulation with bioactive components that might be relevant for food industry. Furthermore, clarifying the beneficial effects of the studied beverages is relevant not only for healthy subjects but also for those with certain disease conditions (i.e., intestinal inflammation diseases), and may contribute to improve their wellbeing and health, with the consequent social and economic benefits.

DESIGN OF THE CLINICAL STUDY:

Single and combined randomized, double-blind, crossover multiple-dose supplementation trial will be carried out with two beverages (250 ml/day): PS-enriched skimmed milk based fruit beverage rich in β-Cx (sham beverage) and a similar skimmed milk based fruit beverage rich in PS and β-Cx supplemented with GOS (active beverage),as diet supplementation in healthy post-menopausal women.

The Clinical study will take place at the Vitamins Unit of the Clinical Biochemistry Service of the Hospital Universitario Puerta de Hierro-Majadahonda (Madrid, Spain).

Sample size assessment:

The sample size was calculated taking into account the results of total PS and cholesterol obtained in a previous clinical trial (no. NCT01074723). From previous assumption we choose the more conservative option to assure detection of a 7% reduction of cholesterol levels in a mild hypercholesterolemic subjects (e.g. 15 mg/dl) with a type I error of 0.05 and a statistical power of 80%. Furthermore, taking into account that 45% of western population might presented some polymorphisms implicated in the cholesterol absorption process, and assuming a drop-out of 10%, the final sample size should included 40 subjects.

Standard Operating procedures:

Two periods of intervention of 6 weeks separated by a wash-out period of 4 weeks.

During the first trial period, 20 subjects daily will consume the active beverage and 20 subjects will consume the sham beverage for 6 weeks, and after a what-out period of 4 weeks, the type of beverage to be consume during other 6 weeks period will be change (two-by-two cross over assignment). All participants receive sham beverage and active beverage B at some point during the trial but in a different order, depending on the group to which they are assigned.

Sample collection (serum and faeces) will be performed before and after each 6 weeks treatment periods.

All subjects should give written consent to participate in the trial.

The participants will be provided with a list of foods and beverage rich in β-Cx to be avoided during the trial period and will be asked not to change its usual diet and physical activity, to record any side effects during the study, and to complete a semi-quantitative Food Frequency Questionnaire (FFQ) at the end of each intervention period. Question on the organoleptic properties of the beverages will also be included.

ELIGIBILITY:
Inclusion Criteria:

* Age (45-65 years), BMI<35 Kg/m2, amenorrhea over 12 months, non-dieting and non-intake of vitamin D, calcium and ω-3 fatty acids and PS or vitamin-enriched foods or supplements or other dietary bioactive components.

Exclusion Criteria:

* Use of vitamins, hormone replacement therapy, fibrates, statins and a weight losing diet, as well as acute inflammation, chronic medication and infection or intercurrent illness capable of affecting the bioavailability or status of the compounds of interest.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Serum levels of β-Cx | 6 weeks
Serum levels of PS | 6 weeks

SECONDARY OUTCOMES:
Serum lipid profile | 6 weeks
C reactive protein, ferritin, calprotectin, alpha-1-antitrypsin, alpha-1-acid | 6 weeks
  Cardiovascular and inflammation risk markers
Beta C-terminal telopeptide (beta-CrossLaps/betaCTx), osteoprotegerin, Parathyroid hormone (PTH), calcium, phosphorus, Alkaline phosphatase | 6 weeks
  Bone markers
Sterol fecal levels | 6 weeks
β-cryptoxanthin fecal levels | 6 weeks
Interleukins | 6 weeks
beta-carotene oxygenase 1 (BCO1), beta-carotene oxygenase 2 (BCO2), scavenger receptor class B type I (SR-BI), NPC1L1, ATP-binding cassette (ABC) transporters G5 and G8 (ABCG5 and ABCG8) genes | 6 weeks
  Intestinal transporters polymorphisms.
Taxonomic profiles of microbial communities by ribosomal RNA (16SrRNA) gene metagenomic studies. Microbiota characterization. | 6 weeks
  Microbiota characterization.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Granado Lorencio, PhD, Principal Investigator — Hospital Universitario Puerta de Hierro-Majadahonda